CLINICAL TRIAL: NCT06203665
Title: Restoration of Pulmonary Compliance After Laparoscopic Gynaecologic Surgery Using a Recruitment Maneuver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panagiota Griva (Other)
Responsible Party: Sponsor-Investigator, Panagiota Griva, Resident Doctor, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 275/27-04-2023
Record Dates: First submitted 2023-12-06; First posted 2024-01-12 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Atelectasis; Compliance, Patient
MeSH Terms: conditions — Pulmonary Atelectasis; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients enrolled in the protocol (Experimental): An alveolar recruitment nameuver will be performed after the release of pneumoperitoneum
  Interventions: Diagnostic Test: Recruitment Maneuver

INTERVENTIONS:
Diagnostic Test: Recruitment Maneuver — The surgery would be performed under general anaesthesia according to the common practice using protective lung ventilation ( Vt= 6 ml /Kg ideal body weight , RR to maintain end-expiratory CO2 35-45 cmH2O and PEEP= 6- 8 cm H20). An incremental and decremental positive end-expiratory pressure alveolar recruitment maneuver would be performed after release of pneumoperitoneum.

SUMMARY:
To investigate the hypothesis that an alveolar recruitment maneuver after the release of pneumoperitoneum would restore the lung compliance to the baseline values after a laparoscopic gynaecologic surgery.

DETAILED DESCRIPTION:
In recent years, laparoscopic surgery is a common minimal invasive technique which ensures the avoidance of prolong hospital stay, long duration surgery, postoperative pain, operation scars. However, laparoscopic surgery has a negative impact on respiratory mechanics because of the pneumoperitoneum, the changes in position and the appliance of positive pressure ventilation. The increase in abdominal pressure as a result of carbon dioxide insufflation and the typical head-down body position have been shown to impair respiratory function. Application of a pneumoperitoneum-induced elevation of intraabdominal pressure elevates the diaphragm and results in a compression of the dependent ventral lung regions. As a consequence, the amount of atelectasis is increased. The insufflation of CO2 reduced respiratory system compliance, and increased peak inspiratory and mean airway pressures. Additionally, changes to the lithotomy and Trendelenburg position during gynaecologic surgery reduce lung compliance by altering the location of intestinal contents and diaphragm. Especially the Trendelenburg position potentiates the effects of abdominal pressure via gravity and relaxation of the diaphragm; thereby, increasing the airway pressure and reducing the functional residual capacity, which results in further changes in the respiratory system. Therefore, we evaluated the effect of an alveolar recruitment maneuver during gynaecologic laparoscopic surgery by determining the changes in lung compliance.

Design: Prospective study. Setting: Operating room of a hospital. Patients: 31 ASA physical status I and II patients scheduled to undergo gynaecologic laparoscopic surgery in the dorsal lithotomy position.

Interventions: The surgery would be performed under general anaesthesia according to the common practice using protective lung ventilation ( Vt= 6 ml /Kg ideal body weight , RR to maintain end-expiratory CO2 35-45 cmH2O and PEEP= 6- 8 cm H20). An incremental and decremental positive end-expiratory pressure alveolar recruitment maneuver would be performed after release of pneumoperitoneum.

Measurements: Respiratory mechanics including dynamic compliance were measured continuously. Respiratory measures were recorded together with arterial blood gases after induction (T1), with the patient placed in the dorsal lithotomy position (T2), 10 and 90 minutes after CO2 insufflation (T3 and T4), immediately after desufflation in the lithotomy and supine positions (T5 and T6), and 10 minutes after a pulmonary recruitment maneuver at the conclusion of surgery (T7).

Inclusion criteria:

* >18 years old patients
* A gynaecologic laparoscopic surgery would be performed
* Duration of the surgery over 90 minutes

Exclusion criteria:

* Chronic Obstructive Lung Disease with FEV1 < 60 of predicted value
* Lung Emphysema
* BMI > 30
* Hemodynamic instability during the operation
* Acute cor pulmonale

ELIGIBILITY:
Inclusion Criteria:

* >18 years old patients
* A gynaecologic laparoscopic surgery would be performed
* Duration of the surgery over 90 minutes

Exclusion Criteria:

* Chronic Obstructive Lung Disease with FEV1 < 60 of predicted value
* Lung Emphysema
* BMI > 30
* Hemodynamic instability during the operation
* Acute cor pulmonle

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Delta (Δ) Compliance (T1 -T7) | intraoperative, after anesthesia induction and after the release of pneumoperitoneum
  The compliance difference between T1 and T7, where T1 denotes the time of induction to anaesthesia and T7 is the release of pneumoperitoneum time.
Delta (Δ) Compliance (T1 -T8) | intraoperative, after anesthesia induction and after the recruitment maneuver
  The compliance difference between T1 and T8, where T8 is the time of the recruitment maneuver.
Delta (Δ) Compliance (T7 -T8) | intraoperative, after the release of pneumoperitoneum and after the recruitment maneuver
  The different compliance between T7 and T8

SECONDARY OUTCOMES:
Compliance (in mL/cmH2O) | intraoperative (T1-T8)
  Compliance of the lungs measured at the following time frames: after anesthesia induction (T1), after dorsal lithotomy position (T2), after Trendelenburg position (T3), 10 and 90 minutes after CO2 insufflation (T4, T5 respectively), after removal of Trendelenburg position (T6), after desufflation (T7), 10 minutes after an alveolar recruitment maneuver (T8).
Pplateau (in cmH2O) | intraoperative (T1-T8)
  end-inspiratory airway pressure measured at the following time frames: after anesthesia induction (T1), after dorsal lithotomy position (T2), after Trendelenburg position (T3), 10 and 90 minutes after CO2 insufflation (T4, T5 respectively), after removal of Trendelenburg position (T6), after desufflation (T7), 10 minutes after an alveolar recruitment maneuver (T8).
MAP (in mmHg) | intraoperative (T1-T8)
  Mean Arterial Pressure measured at the following time frames: after anesthesia induction (T1), after dorsal lithotomy position (T2), after Trendelenburg position (T3), 10 and 90 minutes after CO2 insufflation (T4, T5 respectively), after removal of Trendelenburg position (T6), after desufflation (T7), 10 minutes after an alveolar recruitment maneuver (T8).
Intraoperative administration of vasoactive agents | intraoperative, after alveolar recruitment maneuver
  The dose of the vasoactive agents administrated to maintain a Mean Arterial Pressure > 65mmHg during the alveolar recruitment maneuver

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Athens "Alexandra", Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No